CLINICAL TRIAL: NCT07078292
Title: The Efficacy and Safety of First-line Treatment Combined With Immunotherapy for Advanced Hepatocellular Carcinoma: a Single Center, Real-world Study
Status: Not yet recruiting | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: E20250416
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma (HCC); Real World Study
Keywords: Hepatocellular Carcinoma; Immunotherapy; Real world study
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Immunotherapy combined with bevacizumab ± TACE/HAIC
- immunotherapy combined with TKI ± TACE/HAIC
- immunotherapy combined with immunotherapy ± TACE/HAIC

SUMMARY:
In recent years, immunotherapy represented by PD-1/PD-L1 inhibitors has continuously brought breakthroughs in the treatment of hepatocellular carcinoma and has gradually become the cornerstone of advanced liver cancer treatment. With positive results from the IMbrave-150 study, the combination of atezolizumab and bevacizumab has been approved for first-line treatment of advanced HCC. Subsequently, multiple immune combination therapy regimens were approved one after another, enriching the first-line treatment options for advanced HCC. At present, combination therapy based on immune checkpoint inhibitors has become the mainstream first-line treatment for advanced HCC, and three main treatment modes have been formed: immune combined with bevacizumab, immune combined with TKI, and immune combined with immunity.

Multiple immune combination therapy regimens have shown a flourishing trend in clinical trials, which has brought some thought-provoking issues to the clinical practice of first-line treatment for advanced HCC. On the one hand, the above studies all used sorafenib/lenvatinib monotherapy as a control, lacking a "head to head" comparison. In real-world scenarios, how to choose between different treatment options depends on the judgment of clinical doctors and drug accessibility, lacking support from research data. On the other hand, the ORR of immune combination therapy is between 20% and 40%, and there are still a large number of patients who have initial treatment resistance to the above regimen and cannot achieve satisfactory therapeutic effects. How to accurately predict/identify the response of different populations to different treatment regimens, and then carry out personalized treatment, is also an important issue facing the first-line treatment of advanced HCC. In addition to systemic anti-tumor therapy, local treatment (such as TACE, HAIC, ablation, radiotherapy, etc.) and surgical treatment are also advantageous weapons for treating advanced HCC, complementing systemic treatment to further improve the prognosis of advanced HCC. However, more clinical research evidence is still needed to support the clinical efficacy data of local treatment combined with systemic treatment in the field of advanced HCC treatment.

Based on the above clinical issues, this study intends to retrospectively and prospectively collect advanced HCC patients who receive first-line immunotherapy in our center, explore the effectiveness and safety of combination therapy based on immune checkpoint inhibitors for first-line treatment of advanced hepatocellular carcinoma in the real world, and reveal the advantageous treatment populations of different immunotherapy regimens (immune+bevacizumab, immune+TKI, immune+immune) in the real world, in order to provide some data reference for the first-line treatment population and regimen selection of advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, male or female not limited
* Non resectable HCC patients diagnosed by tissue/cytology or imaging that meets the diagnostic criteria for HCC
* There must be at least one measurable lesion (RECIST 1.1)
* Use immunotherapy combination therapy as first-line treatment, including atezolizumab+bevacizumab, sintilizumab+bevacizumab analogs, carrelizumab+apatinib, lenvatinib+tirelizumab or sintilizumab, with or without local treatment (including but not limited to TACE, HAIC)
* Have not received systematic anti-tumor treatment in the past
* Child Pugh 5-7 points
* ECOG PS 0-1 points
* Prospective cohort requires patients to have at least one imaging tumor evaluation since baseline;

Exclusion Criteria:

* Lack of baseline data and post-treatment imaging data
* With other malignant tumors
* Merge severe cardiovascular diseases and uncontrollable infections
* Existence of any active autoimmune disease or history of autoimmune disease Expected survival period<3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advaced hepatocellular carcinoma patients，BCLC stage B-C；CNLC stage IIA-IIIB
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 months
  Objective response rate

SECONDARY OUTCOMES:
DCR | 6 months
  Disease Control Rate
Conversion surgery rate | 6 months
PFS | 12 months
  Progression free survival
Overall survival (OS) | 24 months
AE | 12 months
  Adverse events